CLINICAL TRIAL: NCT07277374
Title: Comparison of 6-Lead Electrocardiogram (ECG) Device Data With Standard 12-Lead Electrocardiogram (ECG) Data in Individuals With Different Anthropometric Characteristics
Brief Title: Comparison of a Torso-Based Derived 6-Lead Electrocardiogram (ECG) Device With Standard 12-Lead Electrocardiogram (ECG) in Healthy Volunteers
Acronym: T-ECG
Status: Completed | Type: Observational
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sinem Dogruyol, Associate Professor, Haydarpasa Numune Training and Research Hospital
Other Study IDs: HNH-KAEK 2023/KK/193
Record Dates: First submitted 2025-11-26; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: Electrocardiography; 6-lead ECG; 12-lead ECG; Torso ECG; ECG comparison

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer ECG Group: Participants underwent standard 12-lead ECG and torso-based 6-lead ECG in a single session for comparative interval analysis.
  Interventions: Device: Torso-Based 6-Lead ECG Recording

INTERVENTIONS:
Device: Torso-Based 6-Lead ECG Recording — Non-invasive ECG measurement with torso electrode placement for comparison with standard 12-lead ECG.

SUMMARY:
This study aims to compare electrocardiographic interval measurements obtained from a torso-placed six-lead electrocardiogram (ECG) device (torso-derived ECG; T-ECG) with those obtained from a standard 12-lead electrocardiogram (ECG) in healthy adult volunteers. The torso-derived device synthesizes limb-lead signals using electrodes positioned on the thorax, potentially allowing for faster and more practical ECG acquisition in emergency department settings, operating rooms, and prehospital environments.

A total of 24 participants undergo both standard 12-lead ECG recording and torso-derived 6-lead ECG recording during the same study session. Heart rate (HR), PR interval, QRS duration, QT interval, and corrected QT (QTc) values are analyzed using Bland-Altman agreement analysis and correlation testing. The study also evaluates whether anthropometric characteristics-including body mass index (BMI)-influence the compatibility and agreement between the two measurement systems.

DETAILED DESCRIPTION:
This observational, single-center clinical study evaluates the agreement between a torso-based derived six-lead electrocardiogram (ECG) system and a standard 12-lead electrocardiogram (ECG) in healthy adult volunteers. The study is conducted at Haydarpasa Numune Training and Research Hospital following ethics committee approval (Approval No: 2023/193). Volunteers aged 18 to 65 years without known cardiac disease are enrolled.

Each participant undergoes one standard 12-lead ECG recording followed by a torso-based six-lead ECG recording under identical resting conditions. Electrocardiographic measurements include heart rate (HR), RR interval, PR interval, QRS duration, QT interval, and corrected QT (QTc). Anthropometric characteristics-body weight, height, and body mass index (BMI)-are collected to assess whether body composition influences measurement consistency between the two systems.

Primary analysis includes Bland-Altman agreement statistics and correlation testing between ECG modalities. No drug administration, invasive procedure, randomization, or therapeutic intervention is applied. The study involves minimal risk and is limited to non-invasive surface ECG acquisition.

The expected clinical significance is that, if the torso-based ECG demonstrates measurement compatibility with the standard 12-lead ECG, simplified electrode placement may enable faster ECG acquisition in emergency departments, prehospital evaluations, and clinical scenarios in which limb lead placement is impractical.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

No known cardiovascular disease

No arrhythmia, conduction disorder, or ischemic electrocardiogram (ECG) changes at baseline

Willingness to participate and ability to provide written informed consent

Exclusion Criteria:

Known cardiac disease, including coronary artery disease (CAD), arrhythmia, heart failure, or valvular heart disease

Pacemaker rhythm or baseline abnormal electrocardiogram (ECG) findings

Thoracic deformity or prior thoracic surgery that prevents appropriate electrode placement

Unwillingness to participate or inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy adult volunteers without known cardiovascular disease. All participants undergo both standard 12-lead electrocardiogram (ECG) recording and torso-derived 6-lead electrocardiogram (ECG) recording during a single study session. Participants are screened prior to inclusion to ensure the absence of baseline arrhythmia, ischemia, conduction delay, or structural heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
PR Interval Agreement Between Torso-Derived and Standard 12-Lead Electrocardiogram (ECG) | Single-session baseline ECG recording.
  Mean difference in PR interval between torso-derived six-lead electrocardiogram (ECG) and standard 12-lead ECG recordings obtained during the same resting session.
  Single-session baseline ECG recording.
QRS Duration Agreement Between Torso-Derived and Standard 12-Lead Electrocardiogram (ECG) | Single-session baseline ECG recording.
  Mean difference in QRS duration between torso-derived six-lead ECG and standard 12-lead ECG recordings obtained during the same resting session
QT Interval Agreement Between Torso-Derived and Standard 12-Lead Electrocardiogram (ECG) | Single-session baseline ECG recording
  Mean difference in QT interval between torso-derived six-lead ECG and standard 12-lead ECG recordings obtained during the same resting session.
Heart Rate (HR) Agreement Between Torso-Derived and Standard 12-Lead Electrocardiogram (ECG) | Single-session baseline ECG recording.
  Mean difference in heart rate (HR) between torso-derived six-lead ECG and standard 12-lead ECG recordings obtained during the same resting session.

SECONDARY OUTCOMES:
Agreement Between Torso-Derived 6-Lead Electrocardiogram (ECG) and Standard 12-Lead Electrocardiogram (ECG) Measurements | Single-session recording (baseline only)
  Description:
  Comparison of PR interval, QRS duration, QT interval, and heart rate (HR) measurements obtained from torso-derived 6-lead electrocardiogram (ECG) recordings and standard 12-lead electrocardiogram (ECG) recordings to assess measurement concordance.
  Time Frame:
  Single-session recording (baseline only)

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Training and Research Hospital - Emergency Medicine Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset includes only ECG recordings collected from healthy volunteers, and no identifiable patient-level information is stored or retained. Summary results may be shared in publication form, but raw individual-level data will not be publicly available.